CLINICAL TRIAL: NCT05670600
Title: The Effect of Foot and Ankle Exercise on Pain and Quality of Life in Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ülkü Görgülü Polat, Principal Investigator, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Gaziüniversite
Record Dates: First submitted 2022-12-14; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: Diabetic neuropathic pain; exercise; foot and ankle; pain; quality of life
MeSH Terms: conditions — Diabetic Neuropathies; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Experimental research method was used. There is an intervention and control group. While the intervention group was given foot and ankle exercise training, no intervention was given to the control group. The Visual Analog Scale (VAS) of Neuropathic Pain was calculated by another researcher, who applied foot and ankle exercises to both groups before starting the exercise (1st measurement), fourth (2nd measurement) and at the end of the eighth week (3rd measurement). The Impact on Quality of Life Questionnaire (NePIQoL) was administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): The intervention group received training by sending foot and ankle exercise videos to their mobile phones via WhatsApp.
  Interventions: Other: foot and ankle exercise

INTERVENTIONS:
Other: foot and ankle exercise — Foot and Ankle Exercise Phase
  1. Pulling the foot upwards from the ankle
  2. Bending the foot down from the ankle
  3. Spreading the feet like a fan, moving the toes in and out to the right and left
  4. Circle drawing exercise with ankle
  5. Towel folding exercise
  6. Bottle rolling exercise under the feet (The water in the bottle will be warm tap water)

SUMMARY:
The study will be carried out to determine the effect on pain and quality of life between the groups that received and did not receive foot and ankle exercise training.

DETAILED DESCRIPTION:
In the literature, in patients with diabetic neuropathy who received foot and ankle exercise training; It is observed that it reduces the level of pain and increases the quality of life. Foot and ankle exercise training given to the participants improved blood circulation, improved foot-ankle range of motion, increased foot muscle strength and function, improved diabetic neuropathy symptoms, redistributed plantar pressure during movement, improved sensitivity, and was effective in maintaining balance; It is thought that participants can reduce pain and improve their quality of life with foot and ankle exercise training. While there are studies examining the effect of non-pharmacological interventions such as spa treatment and pulse electromagnetic field therapy in patients with diabetic neuropathy in our country, no study has been found examining the effect of foot and ankle exercise training on pain and quality of life in patients with diabetic neuropathic pain. It is thought that the results of the research will be beneficial in symptom management and improve quality of life in addition to pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Having been diagnosed with Type 2 diabetes for at least one year,
* Diagnosed with diabetic peripheral neuropathy for at least 6 months by EMG by a neurologist,
* Individuals with diabetes mellitus with neuropathic pain who score 12 or higher on the S-Lanns (Self-Leeds Assessment of Neuropathic Symptoms and Sign) pain scale,
* Visual Analogue Scale (VAS) value to be at least 1,
* Receiving medical treatment for diabetic neuropathy,
* Did not receive physical therapy and non-pharmacological treatment during the research period,
* Having no physical and mental problems that will prevent communication,
* Having blood glucose meters at home,
* Individuals with smart device use,

Exclusion Criteria:

* Peripheral vascular complications due to diabetes or another etiology,
* Having a history of surgery on the knee, ankle and hip and indication for surgery during the intervention period,
* Those who cannot communicate on the phone (with hearing problems),
* Having nephropathy, retinopathy and diabetic foot,
* Neurological diseases (stroke, cerebrovascular diseases, epilepsy) and serious musculoskeletal problems (rheumatoid arthritis, osteoarthritis)
* Neurocognitive disorder (Alzheimer's disease, dementia),
* Not taking any physical therapy during the intervention period,
* Patients with deep vein thrombosis, femur fractures, surgical conditions, open wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Change in pain level at 4th and 8th weeks compared to baseline. | Two months
  Pain scores of the patients were checked after foot and ankle exercise training. The scale, developed by Price, McGrath, Rafii, and Buckingham, is a measurement tool that evaluates pain severity. The scale is 10 cm long and is graded on a horizontal line (0 = no pain, 10 = most severe pain). The patient is asked to mark a point on this line that corresponds to the intensity of pain he feels. The marked numerical value indicates the severity of the patient's perception of pain. A VAS value of 1 to 4 indicates mild pain, 5-6 indicates moderate pain, and 7-10 indicates severe pain. As scores increase, the level of pain worsens and general health deteriorates.

SECONDARY OUTCOMES:
Effect of neuropathic pain on quality of life at 4 and 8 weeks change from initial state | Two months
  After the interventions, the patient's scores on the effect of neuropathic pain on quality of life are checked. Poole, Murphy, and Nurmka (2009) developed a questionnaire on the impact of neuropathic pain on quality of life. The scale consisting of 42 items; symptoms were divided into 6 subscales under the headings of relationships, psychological, social activity, physical activity, and personal/self care. The results of the questionnaire on the effect of neuropathic pain on the quality of life were calculated by summing the 42-item scores. The total score range is between 42 and 210. The score range for each item is between 1 and 5.

CONTACTS AND LOCATIONS:
Overall Officials: Ülkü Polat, Prof., Principal Investigator — Gazi University; Selin Çiftçi, Principal Investigator — Gazi University
Locations (1):
- Toros Devlet Hastanesi, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
all IPD underlying results in a publication

REFERENCES:
- [Background] Feldman EL, Callaghan BC, Pop-Busui R, Zochodne DW, Wright DE, Bennett DL, Bril V, Russell JW, Viswanathan V. Diabetic neuropathy. Nat Rev Dis Primers. 2019 Jun 13;5(1):41. doi: 10.1038/s41572-019-0092-1. PMID 31197153
- [Background] Hazari A, Maiya AG, Shivashankara KN, Agouris I, Monteiro A, Jadhav R, Kumar S, Shashi Kumar CG, Mayya SS. Kinetics and kinematics of diabetic foot in type 2 diabetes mellitus with and without peripheral neuropathy: a systematic review and meta-analysis. Springerplus. 2016 Oct 19;5(1):1819. doi: 10.1186/s40064-016-3405-9. eCollection 2016. PMID 27812455
- [Background] van Laake-Geelen CCM, Smeets RJEM, Quadflieg SPAB, Kleijnen J, Verbunt JA. The effect of exercise therapy combined with psychological therapy on physical activity and quality of life in patients with painful diabetic neuropathy: a systematic review. Scand J Pain. 2019 Jul 26;19(3):433-439. doi: 10.1515/sjpain-2019-0001. PMID 31112511
- [Background] Degu H, Wondimagegnehu A, Yifru YM, Belachew A. Is health related quality of life influenced by diabetic neuropathic pain among type II diabetes mellitus patients in Ethiopia? PLoS One. 2019 Feb 4;14(2):e0211449. doi: 10.1371/journal.pone.0211449. eCollection 2019. PMID 30716109
- [Background] Boyle J, Eriksson ME, Gribble L, Gouni R, Johnsen S, Coppini DV, Kerr D. Randomized, placebo-controlled comparison of amitriptyline, duloxetine, and pregabalin in patients with chronic diabetic peripheral neuropathic pain: impact on pain, polysomnographic sleep, daytime functioning, and quality of life. Diabetes Care. 2012 Dec;35(12):2451-8. doi: 10.2337/dc12-0656. Epub 2012 Sep 18. PMID 22991449
- [Background] Dermanovic Dobrota V, Hrabac P, Skegro D, Smiljanic R, Dobrota S, Prkacin I, Brkljacic N, Peros K, Tomic M, Lukinovic-Skudar V, Basic Kes V. The impact of neuropathic pain and other comorbidities on the quality of life in patients with diabetes. Health Qual Life Outcomes. 2014 Dec 3;12:171. doi: 10.1186/s12955-014-0171-7. PMID 25468384
- [Background] Francia P, Anichini R, De Bellis A, Seghieri G, Lazzeri R, Paternostro F, Gulisano M. Diabetic foot prevention: the role of exercise therapy in the treatment of limited joint mobility, muscle weakness and reduced gait speed. Ital J Anat Embryol. 2015;120(1):21-32. PMID 26738255
- [Background] Mueller MJ, Tuttle LJ, Lemaster JW, Strube MJ, McGill JB, Hastings MK, Sinacore DR. Weight-bearing versus nonweight-bearing exercise for persons with diabetes and peripheral neuropathy: a randomized controlled trial. Arch Phys Med Rehabil. 2013 May;94(5):829-38. doi: 10.1016/j.apmr.2012.12.015. Epub 2012 Dec 28. PMID 23276801
- [Background] Cerrahoglu L, Kosan U, Sirin TC, Ulusoy A. Range of Motion and Plantar Pressure Evaluation for the Effects of Self-Care Foot Exercises on Diabetic Patients with and Without Neuropathy. J Am Podiatr Med Assoc. 2016 May;106(3):189-200. doi: 10.7547/14-095. PMID 27269974
- [Result] Kluding PM, Pasnoor M, Singh R, Jernigan S, Farmer K, Rucker J, Sharma NK, Wright DE. The effect of exercise on neuropathic symptoms, nerve function, and cutaneous innervation in people with diabetic peripheral neuropathy. J Diabetes Complications. 2012 Sep-Oct;26(5):424-9. doi: 10.1016/j.jdiacomp.2012.05.007. Epub 2012 Jun 18. PMID 22717465
- [Result] Sartor CD, Watari R, Passaro AC, Picon AP, Hasue RH, Sacco IC. Effects of a combined strengthening, stretching and functional training program versus usual-care on gait biomechanics and foot function for diabetic neuropathy: a randomized controlled trial. BMC Musculoskelet Disord. 2012 Mar 19;13:36. doi: 10.1186/1471-2474-13-36. PMID 22429765
- [Result] Ahn S, Song R. Effects of Tai Chi Exercise on glucose control, neuropathy scores, balance, and quality of life in patients with type 2 diabetes and neuropathy. J Altern Complement Med. 2012 Dec;18(12):1172-8. doi: 10.1089/acm.2011.0690. Epub 2012 Sep 17. PMID 22985218
- [Result] Monteiro RL, Sartor CD, Ferreira JSSP, Dantas MGB, Bus SA, Sacco ICN. Protocol for evaluating the effects of a foot-ankle therapeutic exercise program on daily activity, foot-ankle functionality, and biomechanics in people with diabetic polyneuropathy: a randomized controlled trial. BMC Musculoskelet Disord. 2018 Nov 14;19(1):400. doi: 10.1186/s12891-018-2323-0. PMID 30428863
- [Result] Monteiro RL, Ferreira JSSP, Silva EQ, Donini A, Cruvinel-Junior RH, Verissimo JL, Bus SA, Sacco ICN. Feasibility and Preliminary Efficacy of a Foot-Ankle Exercise Program Aiming to Improve Foot-Ankle Functionality and Gait Biomechanics in People with Diabetic Neuropathy: A Randomized Controlled Trial. Sensors (Basel). 2020 Sep 9;20(18):5129. doi: 10.3390/s20185129. PMID 32916792
- [Result] Sartor CD, Hasue RH, Cacciari LP, Butugan MK, Watari R, Passaro AC, Giacomozzi C, Sacco IC. Effects of strengthening, stretching and functional training on foot function in patients with diabetic neuropathy: results of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Apr 27;15:137. doi: 10.1186/1471-2474-15-137. PMID 24767584
- [Result] Kanchanasamut W, Pensri P. Effects of weight-bearing exercise on a mini-trampoline on foot mobility, plantar pressure and sensation of diabetic neuropathic feet; a preliminary study. Diabet Foot Ankle. 2017 Feb 20;8(1):1287239. doi: 10.1080/2000625X.2017.1287239. eCollection 2017. PMID 28326159
- [Result] Win MMTM, Fukai K, Nyunt HH, Linn KZ. Hand and foot exercises for diabetic peripheral neuropathy: A randomized controlled trial. Nurs Health Sci. 2020 Jun;22(2):416-426. doi: 10.1111/nhs.12676. Epub 2019 Dec 26. PMID 31876991
- [Result] Chang CF, Chang CC, Hwang SL, Chen MY. Effects of Buerger Exercise Combined Health-Promoting Program on Peripheral Neurovasculopathy Among Community Residents at High Risk for Diabetic Foot Ulceration. Worldviews Evid Based Nurs. 2015 Jun;12(3):145-53. doi: 10.1111/wvn.12091. Epub 2015 May 11. PMID 25963925
- [Result] van Schie CH. Neuropathy: mobility and quality of life. Diabetes Metab Res Rev. 2008 May-Jun;24 Suppl 1:S45-51. doi: 10.1002/dmrr.856. PMID 18351588
- [Result] Sacco IC, Picon AP, Macedo DO, Butugan MK, Watari R, Sartor CD. Alterations in the lower limb joint moments precede the peripheral neuropathy diagnosis in diabetes patients. Diabetes Technol Ther. 2015 Jun;17(6):405-12. doi: 10.1089/dia.2014.0284. Epub 2015 Feb 9. PMID 25664904